CLINICAL TRIAL: NCT01417221
Title: Renal Sympathetic Modification in Patients With Essential Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Collaborators: Jiangsu Provincial People's Hospital (Other); Zunyi Medical College (Other); Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Yuehui Yin, Director and Professor, Dept. of Cardiology, the second affiliated hospital of Chongqing Medical University, Chongqing Cardiac arrhythmias service center, The Second Affiliated Hospital of Chongqing Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SWAN-HT
Record Dates: First submitted 2011-08-15; First posted 2011-08-16 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Essential Hypertension
Keywords: renal artery; sympathetic nerves; modification; essential hypertension; primary hypertension
MeSH Terms: conditions — Essential Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- renal sympathetic modification (Experimental): Renal artery ablation to modify sympathetic activity in patients with essential hypertension.
  Interventions: Procedure: renal sympathetic modification
- Absolute medicine therapy (No Intervention): Maintenance of anti-hypertensive medications only

INTERVENTIONS:
Procedure: renal sympathetic modification — Device: THERMOCOOL® Catheter Renal sympathetic modification with a catheter-based procedure
  Other Names: renal denervation
  Arms: renal sympathetic modification

SUMMARY:
The purpose of this study is to observe the incident of composite cardiovascular events after renal sympathetic modification using THERMOCOOL® catheter in patients with essential hypertension, and evaluate safety and efficacy of the intervention.

DETAILED DESCRIPTION:
Hypertension is a common cardiovascular disease, and is also an important risk factor for heart-brain-renal diseases, with relatively low controlled rate. Traditional pharmacological therapies are used in clinical practice without breakthrough for long time. Previous studies confirmed that sympathetic nerves activity contributed to development and perpetuation of hypertension. Renal ablation for sympathetic modification is a new method which is proved to be effective in decreasing sympathetic nerves activity. We assume that modifying renal sympathetic activity by ablation is effective and safe in treatment of hypertension. This trial is going to recruit 200 patients (Ablation group VS Control group = 1:1) with a follow-up duration of 3 years. Patients in ablation group will receive additional necessary anti-hypertensive medications besides expectant intervention, and patients in control group will receive appropriate anti-hypertensive medications only. We aim to observe the incident of composite cardiovascular events after renal sympathetic modification using THERMOCOOL® catheter in patients with hypertension, and evaluate safety and efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, and ≤ 75 years old of age
* more than half a year history of hypertension, except for valvular heart disease
* recently at least three times office blood pressure suggest systolic blood pressure of 140mmHg or more and/or a diastolic blood pressure of 90mmHg or more
* estimated glomerular filtration rate (eGFR) of ≥ 45mL/min
* is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

* secondary hypertension
* isolated systolic hypertension
* estimated glomerular filtration rate (eGFR) of < 45mL/min
* has the history of renal restenosis or renal stents implantation
* has experienced AMI (old myocardial infarction is not excluded), unstable angina pectoris, cerebrovascular accidents, and alimentary tract hemorrhage within 3 months
* patients with sick sinus syndrome
* pregnant women
* mental disorders
* patients that have allergy to contrast agent
* patients that do not go with follow-up
* others such as researcher considers it is not appropriate to be included into the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-08 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
composite cardiovascular events | three years
  Comprising myocardial infarction, stroke, heart failure, sudden death

CONTACTS AND LOCATIONS:
Locations (1):
- 2ndChongqingMU, Chongqing, Chongqing Municipality, China